CLINICAL TRIAL: NCT00064688
Title: Genomic Dissection of a QTL Affecting the Lipid Profile
Status: Withdrawn | Type: Observational
Why Stopped: This protocol was created to support work as part of an NIH-funded study.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1230; R01HL074168 (NIH)
Record Dates: First submitted 2003-07-10; First posted 2003-07-14 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemia, Familial Combined
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity; Hyperlipidemia, Familial Combined

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
To search for the genetic cause of the metabolic syndrome, a lipid disorder that poses a major risk for coronary heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

The metabolic syndrome is a common disorder posing a significant major risk for coronary heart disease and early mortality in the Western hemisphere. Central to its cardiovascular complications is the association of the syndrome with the specific abnormalities in plasma lipid and lipoprotein profiles including increased plasma triglycerides, decreased HDL cholesterol, and predominance of dense lipoprotein particles. In search for the genetic etiology of this lipid disorder, the investigators identified a quantitative trait locus (QTL) on human chromosome 7q36 strongly linked to variation in plasma lipid levels. They hypothesize that this QTL contains genetic variants that contribute to alterations in biologic pathways underlying the genesis of the lipid disorder.

DESIGN NARRATIVE:

The study will search for the genetic cause of the metabolic syndrome, a lipid disorder that poses a major risk for coronary heart disease. The investigators have identified a quantitative trait locus (QTL) on human chromosome 7q36 strongly linked to variation in plasma lipid levels. The investigators hypothesize that this QTL contains genetic variants that contribute to alterations in biologic pathways underlying the genesis of the lipid disorder. To test for this hypothesis, they propose a comprehensive approach utilizing established resources and expertise to identify the functional sequence variants within this QTL. Specifically, they will 1.) identify single nucleotide polymorphisms (SNPs) and their haplotype and linkage disequilibrium structure across the entire QTL region; 2.) Analyze association of informative SNPs with plasma triglyceride levels, LDL levels, and lipoprotein density fractions using variance component linkage/disequilibrium analyses; and 3.) Identify potentially functional sequence variants in associated genes or genomic regions using Bayesian quantitative trait nucleotide analysis. This comprehensive application of newly available genomic technologies, novel statistical approaches, the DNA and phenotypic information available, and the consortium of expertise assembled behind this project will ensure the successful elucidation of the genetic etiology of this lipid disorder and consequently the development of effective means for prevention and/or treatment of cardiovascular complications of the metabolic syndrome.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)